CLINICAL TRIAL: NCT06011837
Title: Effects of Altered Auditory Feedback on Speech Fluency
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1906848293
Record Dates: First submitted 2023-05-09; First posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Stuttering, Adult
MeSH Terms: conditions — Stuttering

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Altered Auditory Feedback (Experimental): Participants in this arm will use the Mumble Melody application over the course of 1 month
  Interventions: Device: Altered Auditory Feedback

INTERVENTIONS:
Device: Altered Auditory Feedback — Mumble Melody is an application that leverages Altered Auditory Feedback (AAF). During AAF, a person's speech is altered in near-real time. Mumble Melody modulates the user's voice and plays it back to them while they are speaking. Included are Unaltered (raw voice), Whisper (voiceless sound), Reverb (cathedral sound), and Harmonized (robotic sound) voice transformations.
  Other Names: Musically Modulated Auditory Feedback; Mumble Melody

SUMMARY:
The purpose of the study is to use altered auditory vocal feedback to increase fluency in people who stutter and to examine changes in this effect over the course of a one month period occurring outside the laboratory setting.

DETAILED DESCRIPTION:
The Mumble Melody app applies voice transformations (or "modes") to a user's voice in real-time while they are speaking. The modes include Unaltered, Whisper, Reverberated, and Harmonious voice transformations. The Mumble Melody Longitudinal Study is a month-long online study in which we will be investigating the longer term effects of using the Mumble Melody app for people who stutter. During the course of a month, eligible participants will use the Mumble Melody app daily for however long, on whichever modes, and in whichever settings they wish. Additionally, we will be sending an online platform for participants to conduct weekly at-home testing sessions, in which they will be asked to record their voice during various speech tasks, both with and without the Mumble Melody app. During testing sessions, we will collect voice recordings from participants.

Step 1: Participants will sign a consent form via Redcap. Participants will need an Apple device compatible with the Mumble Melody app.

Step 2: Participants will receive an additional form via Redcap through which they can input information about what device they will be using for the Mumble Melody study, as well as shipping information to receive wired headphones and a headphone jack (which are necessary to use the app).

Step 3: Participants conduct an initial screening session through an online platform, in which they respond to 3 90-second open questions and conduct a passage reading task. We will be collecting voice recordings as they speak within the sessions.

Step 4: Participants' eligibility will be determined using the voice recordings received from step 3. The amount of stuttering-like events and total number of syllables within the recordings will determine if participants have a moderate to severe stutter, meaning they will be eligible for the study.

Step 5: Eligible participants are shipped wired headphones and a headphone jack adapter

Step 6: Participants will fill out an initial survey and optional OASES (Overall Assessment of the Speaker's Experience of Stuttering) assessment of through an online platform.

Step 7: Participants conduct a baseline testing session. During this testing session, participants will answer survey questions, record answers to 2 90-second open response questions without using the Mumble Melody app, follow a step-by-step guide to download and set up the Mumble Melody app, record answers to 2 90-second open response for each of the 4 modes on the Mumble Melody app, and finally record answers to 2 90-second open response questions without using the Mumble Melody app.

Step 8: Step 8: For the following 28 days, participants will be told to use the app as they wish. We will collect app usage logs, which provide timestamps indicating which mode was used and length of use. Participants will receive an additional monetary reward if they use the app for at least 5 minutes for 4 out of 6 days each week.

Step 9: Participants conduct 4 testing sessions, one at the end of each week of the study (day 8, 15, 22, and 29). During each testing session, participants will answer survey questions, record answers to 2 90-second open response questions without using the Mumble Melody app, record answers to 2 90-second open response for each of the 4 modes on the Mumble Melody app, and finally record answers to 2 90-second open response questions without using the Mumble Melody app.

Step 10: After the study, participants will be sent a final survey asking questions on their experience throughout the study and their feedback for the app.

ELIGIBILITY:
Inclusion Criteria:

* Identifies as a person who stutters
* Is US citizen or green card holder currently residing in the US
* Has one of the following Apple devices:
* iPhone with iOS 12.0 or later
* iPad with iPadOS 12.0 or later
* iPod touch with iOS 12.0 or later
* Mac with macOS 11.0 or later and an Apple M1 chip or later
* Has a SEPARATE browser-supporting device with a microphone
* Is able to conduct the study in English
* Qualifies based on an initial screening evaluation (Greater than 2.5% Stuttering-Like Dysfluencies per syllable)

Exclusion Criteria:

-

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-05-26 (Actual); Primary Completion 2024-07-14 (Estimated); Study Completion 2024-07-14 (Estimated)

PRIMARY OUTCOMES:
Significant change in fluency in one of four modes (Unaltered, Whisper, Reverb, Harmonize) between the baseline testing session and the end of week 4. | Calculated at the end of the study for time points 1-week, 2-weeks, 3-weeks, and 4-weeks
  Fluency change From Baseline - Week 4 Measured by Stuttering-Like Dysfluencies within voice recordings from participants

SECONDARY OUTCOMES:
Frequency of Mode Usage | Calculated every day for 4 weeks
  Number of times participants use each modes per day throughout the study
Duration of Mode Usage | Calculated every day for 4 weeks
  Length of times participants use different modes per day throughout the study
Survey data on experience using the application | immediately after the intervention
  A final survey provided for participants' feedback on their experience
Significant change in fluency in one of four modes (Unaltered, Whisper, Reverb, Harmonize) between the baseline testing session and end of week 1, 2, and 3. | Calculated at the end of the study for time points: Baseline, 1-week, 2-weeks, 3-weeks, and 4-weeks
  Fluency change From Baseline - Week 1,2,3 Measured by Stuttering-Like Dysfluencies within voice recordings from participants
Significant change in fluency in the Baseline (No Auditory Feedback) condition between baseline and end of week 1, 2, 3, and 4. | Calculated at the end of the study for time points: Baseline, 1-week, 2-weeks, 3-weeks, and 4-weeks
  Fluency change From Baseline - Week 1,2,3,4 Measured by Stuttering-Like Dysfluencies within voice recordings from participants
Significant change in fluency in the Final (No Auditory Feedback) condition between baseline and end of week 1, 2, 3, and 4. | Calculated at the end of the study for time points: Baseline, 1-week, 2-weeks, 3-weeks, and 4-weeks
  Fluency change From Baseline - Week 1,2,3,4 Measured by Stuttering-Like Dysfluencies within voice recordings from participants
Significant change in fluency for the Final (No Auditory Feedback) condition in comparison to the baseline (No Auditory Feedback) condition, for each testing session | Calculated at the end of the study for time points: Baseline, 1-week, 2-weeks, 3-weeks, and 4-weeks
  Fluency change From Baseline (No Auditory Feedback) - Final (No Auditory Feedback) for each Testing Session Measured by Stuttering-Like Dysfluencies within voice recordings from participants
Significant change in fluency for each mode in comparison to the baseline (No Auditory Feedback) condition, for each testing session | Calculated at the end of the study for time points: Baseline, 1-week, 2-weeks, 3-weeks, and 4-weeks
  Fluency change From Baseline (No Auditory Feedback) - each Mode for each Testing Session Measured by Stuttering-Like Dysfluencies within voice recordings from participants
Significant change in fluency for each non- control mode (Whisper, Reverb, Harmonize) in comparison to the control mode (Unaltered), for each testing session | Calculated at the end of the study for time points: Baseline, 1-week, 2-weeks, 3-weeks, and 4-weeks
  Fluency change From Unaltered Mode - Whisper/Reverb/Harmonize modes for each Testing Session Measured by Stuttering-Like Dysfluencies within voice recordings from participants

CONTACTS AND LOCATIONS:
Overall Officials: Satrajit Ghosh, PhD, Principal Investigator — Massachusetts Institute of Technology
Locations (1):
- Massachusetts Institute of Technology, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Subjects can choose to consent to having their audio recordings and survey answers shared with the researchers of this study and other qualified researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting September 2024
Access Criteria: The data will be shared through an online repository such as Dataverse, with associated data use agreement to not use the information to identify participants, and to reuse the data in a manner to verify the outcomes of the research or related research. Based on our consent form, individual data may also be submitted to databases for any broad reuse.

DOCUMENTS (3):
  • Study Protocol (2023-05-01): https://cdn.clinicaltrials.gov/large-docs/37/NCT06011837/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-01): https://cdn.clinicaltrials.gov/large-docs/37/NCT06011837/SAP_001.pdf
  • Informed Consent Form (2023-05-01): https://cdn.clinicaltrials.gov/large-docs/37/NCT06011837/ICF_002.pdf